CLINICAL TRIAL: NCT00164632
Title: California No More Falls! Senior Injury Prevention Program
Brief Title: No More Falls Injury Prevention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCIPC-3339; U17/CCU918906
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Falls
MeSH Terms: interventions — Counseling; Exercise; Referral and Consultation

INTERVENTIONS:
Behavioral: counselling, exercise, referrals (behavior)

SUMMARY:
A randomized controlled multi-component fall prevention study for older adults. The study integrates fall prevention into an existing community-based public health program for older adults.

DETAILED DESCRIPTION:
A randomized controlled multi-component fall prevention study for older adults. The study integrates fall prevention into an existing community-based public health program for older adults. The study will evaluate the effectiveness of a fall prevention intervention among 552 seniors attending Preventive Health Care for the Aging (PHCA) clinics in two counties: urban San Diego county and rural Humboldt county. The intervention includes four elements: education about fall risk factors, referrals to community exercise programs to increase strength and balance, medication review, and home modification to reduce home hazards. The goal of the intervention is to reduce incidence of falls requiring hospitalization by 10%. Results of the study, which are expected to be completed by October 2004, will help guide future efforts to develop multifaceted fall prevention programs.

ELIGIBILITY:
Inclusion Criteria: PHCA clients age 65+ -

Exclusion Criteria: Age <65

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 552
Dates: Start 2001-10

PRIMARY OUTCOMES:
Number of falls reported after 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Barb Alberson, MPH, Principal Investigator — California Department of Health Services